CLINICAL TRIAL: NCT02092818
Title: EXPERT, EXPosurE Registry RiociguaT in Patients With Pulmonary Hypertension
Acronym: EXPERT
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16657; AD1301 (Other: company internal)
Record Dates: First submitted 2014-03-19; First posted 2014-03-20 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — riociguat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Patients who have been prescribed Adempas for a medically appropriate use
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) — The decision on clinical management of the patient including the actual treatment duration will be determined solely by the physician not by the clinical study protocol (CSP)

SUMMARY:
In accordance with the regulatory guidance this registry has been designed to collect information about the long-term safety of Adempas in real clinical practice outside the regulated environment of a controlled clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients who start or are on treatment with Adempas
* Written informed consent

Exclusion Criteria:

* Patients currently participating in an interventional clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been prescribed Adempas® for a medically appropriate use
Sampling Method: Probability Sample
Enrollment: 1316 (Actual)
Dates: Start 2014-05-31 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Up to 4 years
Number of serious adverse events | Up to 4 years
All-cause mortality | Up to 4 years

SECONDARY OUTCOMES:
Number of adverse event (AE) in the different pulmonary hypertension(PH) indications (pulmonary arterial hypertension (PAH) chronic thromboembolic pulmonary hypertension(CTEPH) | Up to 4 years
Number of serious adverse event (SAE) in different PH indications (PAH and CTEPH) | Up to 4 years
Incidence of AE of special interest overall | Up to 4 years
Incidence of AE of special interest in different PH indications (PAH, CTEPH) | Up to 4 years
6 minute walking distance | Up to 4 years
Functional class of pulmonary hypertension according to NYHA/ WHO | Up to 4 years
  NYHA/ WHO: New York Heart Association / World Health Organization
Borg Dyspnoea Index | Up to 4 years
EQ5D visual analogue scale (VAS) score | Up to 4 years
  EQ5D: EurQuol 5 dimensions (questionnaire)
Number of patients with hemodynamic measurements | Up to 4 years
Concentration of biomarkers for heart insufficiency (Brain Natriuretic Peptide (BNP) and N-Terminal pro BNP (NTpro BNP)) | Up to 4 years
Number of hospitalization | Up to 4 years
Number of outpatient visits | Up to 4 years
Number of days in home care | Up to 4 years
Number of days in rehabilitation | Up to 4 years
Number of days in nursery home | Up to 4 years
Drug treatment for PH | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (28):
- Multiple Locations, Argentina
- Multiple Locations, Australia
- Multiple Locations, Austria
- Multiple Locations, Belgium
- Multiple Locations, Canada
- Multiple Locations, Colombia
- Multiple Locations, Czechia
- Multiple Locations, Denmark
- Multiple Locations, Estonia
- Multiple Locations, Finland
- Multiple Locations, France
- Multiple Locations, Germany
- Multiple Locations, Greece
- Multiple Locations, Ireland
- Multiple Locations, Italy
- Multiple Locations, Luxembourg
- Multiple Locations, Netherlands
- Multiple Locations, Norway
- Multiple Locations, Portugal
- Multiple Locations, Russia
- Multiple Locations, Saudi Arabia
- Multiple Locations, Slovakia
- Multiple Locations, Spain
- Multiple Locations, Sweden
- Multiple Locations, Switzerland
- Multiple Locations, Taiwan
- Multiple Locations, Turkey (Türkiye)
- Multiple Locations, United Kingdom